CLINICAL TRIAL: NCT02136212
Title: Positive Emotional Processing: Exploring Novel Treatment Targets in Social Phobia - New Data
Brief Title: Positive Emotional Processing: Exploring Novel Treatment Targets in Social Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Charles Taylor, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R00MH090243 (NIH); R00MH090243 (NIH)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Approach-positive AAT (Experimental): Participants will receive 4 sessions over 2 weeks of a computerized AAT procedure designed to increase automatic approach responses for positive social cues.
  Interventions: Behavioral: Approach-positive AAT
- Control AAT (Placebo Comparator): Participants will receive 4 sessions over 2 weeks of a computerized AAT procedure in which there is no contingency between arm movement and positive social cues.
  Interventions: Behavioral: Control AAT

INTERVENTIONS:
Behavioral: Approach-positive AAT
  Arms: Approach-positive AAT
Behavioral: Control AAT
  Arms: Control AAT

SUMMARY:
The purpose of this study is to test the effects of a computerized approach/avoidance training (AAT) procedure in a sample of individuals diagnosed with social anxiety disorder (SAD). The training procedure is designed to modify automatic approach responses for positive social stimuli. Previous research has shown that a single administration of approach-positive AAT influences social behavior in the laboratory. The goal of this study is to examine the effects of a four-session AAT procedure on measures of positive social-emotional functioning. The investigators hypothesize that individuals assigned to the approach-positive AAT condition will demonstrate larger increases in positive affect and improvements in social relationship functioning from pre- to post-assessment compared to those assigned to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Principal psychiatric diagnosis of generalized social anxiety disorder
* Liebowitz Social Anxiety Scale (LSAS) score ≥ 60
* Ability to read and speak English sufficiently to complete study procedures

Exclusion Criteria:

* History of psychosis, mania, or substance dependence
* Current severe medical disorder that requires inpatient treatment or frequent medical follow ups including but not limited to: unstable hypertension, unstable angina, unstable diabetes mellitus, unstable cardiac arrhythmias, transient ischemic attacks, severe coronary artery disease, severe peripheral vascular disease, severe hepato-gastro-intestinal disease, severe infectious disease (e.g. HIV), recurrent severe headache or migraine, fainting spells, seizures, and history of traumatic brain injury with loss of consciousness >30 minutes
* Current use of the following medications: antidepressants, benzodiazepines, antipsychotics, mood stabilizers, or other drugs that can acutely affect the hemodynamic response (methylphenidate and acetazolamide)
* Caffeine intake >10 cups/day or recent significant changes in consumption
* MRI exclusions, including claustrophobia, cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a metal worker/welder, history of eye surgery/eyes washed out because of metal, women who are or may be pregnant (determined by a positive pregnancy test), women using an intrauterine device, vision problems uncorrectable with lenses, claustrophobia, inability to lie still on one's back for 60 minutes; prior neurosurgery; older tattoos with metal dyes; unwillingness to remove nose, ear, tongue, or face rings.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in positive affect (Positive and Negative Affect Schedule) | 1 month
  Change from pre- to post-assessment in positive affect.
Change from baseline in social connectedness (Social Connectedness Scale - Revised) | 1 month
  Change from pre- to post-assessment in social connectedness.

SECONDARY OUTCOMES:
Change from baseline in social relationship functioning (Interpersonal Outcomes Scale) | 1 month
  Change from pre- to post-assessment in frequency of social approach behaviors and relationship satisfaction.
Change from baseline in social anxiety symptoms (Liebowitz Social Anxiety Scale) | 1 month
  Change from pre- to post-assessment in social anxiety symptoms.

OTHER OUTCOMES:
Change from baseline in blood oxygen level dependent (BOLD) response in the striatum, amygdala, and medial prefrontal cortex, as measured with functional magnetic resonance imaging (fMRI) | 1 month
  Change from pre- to post-assessment in neural activation during social reward processing.
Change from baseline in social anxiety disorder (SAD) related psychopathology, including depression and anhedonia. | 1 month
  Change from pre- to post-assessment in symptoms of depression and anhedonia

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Taylor, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego; Psychiatry Clinical Research, San Diego, California, United States

REFERENCES:
- [Derived] Hunt C, Caudle MM, Paulus MP, Stein MB, Taylor CT, Bomyea J. Reduced neural activation during positive social approach is associated with better response to approach avoidance training for social anxiety disorder. J Mood Anxiety Disord. 2025 Feb 7;10:100110. doi: 10.1016/j.xjmad.2025.100110. eCollection 2025 Jun. PMID 40657593
- [Derived] Bomyea J, Sweet A, Davey DK, Boland M, Paulus MP, Stein MB, Taylor CT. Randomized controlled trial of computerized approach/avoidance training in social anxiety disorder: Neural and symptom outcomes. J Affect Disord. 2023 Mar 1;324:36-45. doi: 10.1016/j.jad.2022.12.054. Epub 2022 Dec 19. PMID 36549342